CLINICAL TRIAL: NCT03415893
Title: High-resolution Esophageal Manometry in Teenagers With Esophageal Atresia
Brief Title: High-resolution Esophageal Manometry
Status: Completed | Type: Observational
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, CECILIA CURVALE, PI, Hospital El Cruce
Other Study IDs: High-resolution manometry
Record Dates: First submitted 2018-01-22; First posted 2018-01-30 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Atresia
Keywords: high-resolution manometry; esophageal atresia; teenagers
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
EA is one of the most frequent birth defects, with an incidence of 1 in 3000 live births1. Until the 1950s, these patients had 100% mortality; nowadays, the survival rate is greater than 90%, and only those with associated severe malformations die1-5.

Type C EA (atresia of the esophageal proximal segment with tracheoesophageal fistula between the trachea and the distal segment) is the most common variant, since it is present in 85% of the cases6-8. There is evidence that the esophageal motor disorder present in these children is secondary to a congenital neuromuscular disorder and a postoperative disorder9-14. Patients that survive the operation have greater risk of developing gastroesophageal reflux disease (GERD), caused by anomalies in the esophageal motility and its resulting delay in the evacuation of acid of the esophageal lumen.

There was a hypothesis that suggested that motility alteration could contribute to dysphagia and to the high prevalence of gastroesophageal reflux in these patients15-18. Also, there were reports of a greater incidence of severe esophagitis with requirement of fundoplication, which shows a larger failure rate17-18. Esophageal dysmotility has been proved in children with EA through performance of conventional perfusion manometry.

Lemoine C et al described three motility alteration patterns with HRM in children with repaired EA. Said study allowed a more precise knowledge of segmental esophageal motility19. Currently, there are no reports exclusively made about teenagers with repaired EA that describe segmental esophageal motility with HRM.

ELIGIBILITY:
Inclusion Criteria:

teenagers of more than 12 years old, with repaired EA, orally fed during the last 6 months, with no history of esophageal blockage or dilations, who underwent a HREM

Exclusion Criteria:

* patients under 12 years old

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: teenagers with esophageal atresia and surgically repaired
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Patterns of High Resolution Manometry in teenagers with esophageal atresia | one day
  Number of patients with patterns of complete aperistalsis, pressurization and distal esophageal contraction in High Resolution Manometry

CONTACTS AND LOCATIONS:
Overall Officials: cecilia curvale, Principal Investigator — Hospital El Cruce
Locations (1):
- Hospital El Cruce, San Juan Bautista, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No